CLINICAL TRIAL: NCT03895840
Title: The Effect of Intra-articular Bilateral Knee Injections of Zilretta on Osteoarthritis Research Society International (OARSI) Recommended Physical Performance Measures in Adults With Knee Osteoarthritis
Brief Title: The Effect of Intra-articular Bilateral Knee Injections of Zilretta on Performance Measures in Adults With Knee OA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00142926
Record Dates: First submitted 2019-03-25; First posted 2019-03-29 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Triamcinolone; FX006

STUDY DESIGN:
Intervention Model Description: This will be an open-label study to determine the functional effects of IA injection of Zilretta into bilateral knees of 70 subjects with KL grade 2-4 symptomatic knee OA. Measurement of OARSI recommended physical performance measures, patient-reported physical function, quality of life and pain at baseline, 6, 12 and 24 weeks will allow assessment of short and long-term effects, consistent with OARSI and OMERACT recommendations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intra-articular Zilretta injection (Experimental): 32 mg Zilretta in a 5ml diluent for each knee, per manufacturer guidelines
  Interventions: Drug: Zilretta

INTERVENTIONS:
Drug: Zilretta — Zilretta (triamcinolone acetonide extended-release injectable suspension) is indicated as an intra-articular injection for the management of pain due to knee osteoarthritis.
  Other Names: FX006; Triamcinolone acetonide extended-release

SUMMARY:
This study will be an open-label trial to determine the functional effects of bilateral IA injections of Zilretta into knee joints of 70 subjects with bilateral KL grade 2-4 symptomatic knee osteoarthritis (OA). Measurement and evaluation of outcomes at baseline, 6, 12 and 24 weeks will allow assessment of short and long-term effects, consistent with Osteoarthritis Research Society International (OARSI) and Outcome Measures in Rheumatology (OMERACT) recommendations.

DETAILED DESCRIPTION:
The primary aim of the proposed study is to demonstrate the effect of IA injection of Zilretta on physical performance measures in adults with bilateral knee OA. The primary study endpoint will be the change in OARSI recommended physical performance tests (30-second chair standing test, 40m fast-paced walking test, stair ascent) 12 weeks after treatment.

The secondary outcome will be the change in Knee Injury and Osteoarthritis Outcome Score (KOOS-PS) patient-reported physical function short form.

The tertiary outcomes will be the change in KOOS-Quality of life subscale (QoL) and Numerical Rating Scale (NRS) for pain. All outcomes will be assessed at 6- and 24-week follow-up as well to define the course and trajectory of effects.

Specific Aim 1: To determine the extent to which intra-articular (IA) injection of Zilretta in patients with bilateral knee OA improves physical performance (OARSI recommended physical performance measures).

Primary Hypothesis 1: Bilateral knee intra-articular injection of Zilretta results in improved physical performance detectable at 6 weeks, 12 weeks (primary), and 24 weeks.

Specific Aim 2: To determine the extent to which IA injection of Zilretta in patients with bilateral knee OA improves physical function (KOOS-PF).

Hypothesis 2: Bilateral knee IA injection of Zilretta results in improved patient-reported physical function (KOOS-PS) at 6 weeks,12 weeks (primary), and 24 weeks.

Specific Aim 3: To determine the extent to which bilateral knee IA injection of Zilretta in patients with bilateral knee OA improves quality of life (KOOS-QoL).

Hypothesis 3: Intra-articular (IA) bilateral knee injection of Zilretta in patients with bilateral knee osteoarthritis results in improved quality of life (KOOS-QoL) detectable at 6 weeks, 12 weeks (primary), and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 30 years or older with symptomatic bilateral knee OA
* Symptomatic knee OA will be defined as the presence of a definite osteophyte or joint space narrowing (KL Grade ≥2) on posteroanterior (PA) fixed flexion knee radiographs in subjects limited by bilateral pain rated on a Numerical Rating Scale as ≥ 4/10 on more than half of the days over the past month. Radiographic change must be visible at standard image size, irrespective of capability to detect more subtle changes through digital enhancement.
* Bilateral knee symptoms for ≥ 3 months prior to screening
* Has undergone at least one prior conservative osteoarthritis treatment (e.g. Physical therapy, analgesics)
* Body Mass Index ≤ 41 kg/m2
* Ambulatory
* Willing and able to comply with the study procedures and visit schedules and ability to follow verbal and written instructions.
* Willingness to abstain from the use of protocol-restricted medications during the study after signing informed consent and also willing to abstain from use of all analgesics other than acetaminophen 1 week prior to beginning of treatment.

Exclusion Criteria:

* Current consumption of more than 14 alcoholic drinks per week
* Clinical signs and symptoms of active knee infection or crystal disease of either knee within 1 month of screening
* Diagnosed with rheumatoid arthritis, Reiter's syndrome, psoriatic arthritis, gout, ankylosing spondylitis, or arthritis secondary to other inflammatory diseases; HIV, viral hepatitis; chondrocalcinosis, Paget's disease, or villonodular synovitis
* Diagnosed with leukemia, known presence of metastatic malignant cells, or ongoing or planned chemotherapeutic treatment.
* A gout attack in the past 2 years.
* Diseases of the spine, hip or other lower extremity joints judged by the investigator to be contributing to the pain in either knee (i.e. sciatica, nerve pain, hip OA). Note: Patients with hip replacement in either hip may be enrolled provided there is sufficient pain relief after hip replacement that analgesics are not required.
* Untreated symptomatic injury of either knee (e.g., acute traumatic injury, anterior cruciate ligament injury, clinically symptomatic meniscus injury characterized by a mechanical issue such as locking or catching).
* Uncontrolled diabetes (HbA1c >7.2)
* Women who report pregnancy or childbearing potential and not using acceptable contraceptive measures (oral contraceptive, long acting reversible contraceptive therapy) (due to the potential for change in body mass and distribution to alter knee symptoms over the period of follow-up).
* Presence of surgical hardware or other foreign body intended to treat arthritis or cartilage-related pathology in either knee.
* Arthroscopy or open surgery of either knee within 6 months of screening.
* Planned/anticipated surgery of either knee during the study period.
* Use of systemic immunosuppressant within 6 weeks of screening.
* Oral corticosteroids (investigational or marketed) within 2 weeks of screening (unless on chronic stable dose for >3 months).
* IA corticosteroid (investigational or marketed) in either knee within 3 months of screening.
* IV or IM (Intramuscular) Corticosteroid injection (investigational or marketed) within 3 months of screening.
* Any other IA drug/biologic use within 6 months of screening or 5 half-lives (whichever is longer) (e.g., hyaluronic acid, platelet-rich plasma (PRP) injection, stem cells, prolotherapy and amniotic fluid injection).
* Any documented clinically significant degree of cognitive impairment or other condition, finding, or psychiatric illness at screening which, in the opinion of the investigator, could compromise subject safety.
* Any condition other than OA of the knee which, in the opinion of the investigator, affects the ability to ambulate to a sufficient degree to interfere with the assessment of the safety and treatment effects of the study injection.
* Participated in any interventional drug or device trial within 30 days prior to screening or concurrent participation in another research study that could complicate interpretation of the study findings.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neil A Segal, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Maricar N, Callaghan MJ, Felson DT, O'Neill TW. Predictors of response to intra-articular steroid injections in knee osteoarthritis--a systematic review. Rheumatology (Oxford). 2013 Jun;52(6):1022-32. doi: 10.1093/rheumatology/kes368. Epub 2012 Dec 22. PMID 23264554
- [Background] Murray CJ, Vos T, Lozano R, Naghavi M, Flaxman AD, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gonzalez-Medina D, Gosselin R, Grainger R, Grant B, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Laden F, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Levinson D, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mock C, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiebe N, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, AlMazroa MA, Memish ZA. Disability-adjusted life years (DALYs) for 291 diseases and injuries in 21 regions, 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2197-223. doi: 10.1016/S0140-6736(12)61689-4. PMID 23245608
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence of disabilities and associated health conditions among adults--United States, 1999. MMWR Morb Mortal Wkly Rep. 2001 Feb 23;50(7):120-5. PMID 11393491
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and most common causes of disability among adults--United States, 2005. MMWR Morb Mortal Wkly Rep. 2009 May 1;58(16):421-6. PMID 19407734
- [Background] Kraus VB, Conaghan PG, Aazami HA, Mehra P, Kivitz AJ, Lufkin J, Hauben J, Johnson JR, Bodick N. Synovial and systemic pharmacokinetics (PK) of triamcinolone acetonide (TA) following intra-articular (IA) injection of an extended-release microsphere-based formulation (FX006) or standard crystalline suspension in patients with knee osteoarthritis (OA). Osteoarthritis Cartilage. 2018 Jan;26(1):34-42. doi: 10.1016/j.joca.2017.10.003. Epub 2017 Oct 9. PMID 29024802
- [Background] Bodick N, Lufkin J, Willwerth C, Kumar A, Bolognese J, Schoonmaker C, Ballal R, Hunter D, Clayman M. An intra-articular, extended-release formulation of triamcinolone acetonide prolongs and amplifies analgesic effect in patients with osteoarthritis of the knee: a randomized clinical trial. J Bone Joint Surg Am. 2015 Jun 3;97(11):877-88. doi: 10.2106/JBJS.N.00918. PMID 26041848
- [Background] McAlindon TE, Driban JB, Henrotin Y, Hunter DJ, Jiang GL, Skou ST, Wang S, Schnitzer T. OARSI Clinical Trials Recommendations: Design, conduct, and reporting of clinical trials for knee osteoarthritis. Osteoarthritis Cartilage. 2015 May;23(5):747-60. doi: 10.1016/j.joca.2015.03.005. PMID 25952346
- [Background] Dobson F, Hinman RS, Hall M, Marshall CJ, Sayer T, Anderson C, Newcomb N, Stratford PW, Bennell KL. Reliability and measurement error of the Osteoarthritis Research Society International (OARSI) recommended performance-based tests of physical function in people with hip and knee osteoarthritis. Osteoarthritis Cartilage. 2017 Nov;25(11):1792-1796. doi: 10.1016/j.joca.2017.06.006. Epub 2017 Jun 22. PMID 28647467
- [Background] Davis AM, Perruccio AV, Canizares M, Hawker GA, Roos EM, Maillefert JF, Lohmander LS. Comparative, validity and responsiveness of the HOOS-PS and KOOS-PS to the WOMAC physical function subscale in total joint replacement for osteoarthritis. Osteoarthritis Cartilage. 2009 Jul;17(7):843-7. doi: 10.1016/j.joca.2009.01.005. Epub 2009 Jan 31. PMID 19215728
- [Background] Gandek B, Ware JE Jr. Validity and Responsiveness of the Knee Injury and Osteoarthritis Outcome Score: A Comparative Study Among Total Knee Replacement Patients. Arthritis Care Res (Hoboken). 2017 Jun;69(6):817-825. doi: 10.1002/acr.23193. Epub 2017 May 8. PMID 28085998
- [Background] P. Conaghan, V. Strand, D. Hunter. An intra-articular, extended release formulation of triamcinolone (FX006) affords clinically relevant improvements in pain and function of knee osteoarthritis: post-hoc pooled analyses of 3 randomized controlled trials. Osteoarthritis and Cartilage April 2017,Volume 25, Supplement 1, Pages S432-S433

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intra-articular Zilretta Injection
Started | 70
6-Week Follow-Up | 70
12-Week Follow-Up | 65
24-Week Follow-Up | 49
Completed (Primary outcome measures were a priori defined at the 12-week follow-up, while 24-week measurements were included for extended follow-up) | 49
Not Completed | 21
Not completed — Withdrawal by Subject | 21

BASELINE CHARACTERISTICS:
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 70
BMI [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (5.7)
Chair Stand (#) [Mean (Standard Deviation); unit: stands] — The 30 second Chair Standing Test is one of three Osteoarthritis Research Society International (OARSI) recommended minimal core set of performance-based outcome measures in OA research and clinical practice.In this test, the subject will stand up completely from the sitting position so hips and knees are fully extended, then completely back in the seated position. This will be repeated for 30 seconds and the total number of chair stands will be recorded (up and down equals one stand).
  stands | 7.7 (3.6)
Stair Climb (sec) [Mean (Standard Deviation); unit: seconds] — The stair climb test is one of the three Osteoarthritis Research Society International recommended minimal core set of performance-based outcome measures in OA research and clinical practice. The subject will be timed while ascending and descending 9 steps of stairs.
  seconds | 22.1 (28.9)
40m Walk Time (sec) [Mean (Standard Deviation); unit: seconds] — The 40-meter fast paced walk test is one of the three Osteoarthritis Research Society International recommended minimal core set of performance-based outcome measures in OA research and clinical practice.The subjects will be timed to complete a 40 m track course.
  seconds | 37.3 (26.0)
Physical Function (KOOS) [Mean (Standard Deviation); unit: score on a scale] — KOOS-Physical Function (KOOS-PS) Short Form is a parsimonious measure of physical function derived from the KOOS, which is a self-reported outcome score. The KOOS-Physical Function Short Form ranges from 0 to 100 where higher values represents a worse outcome.
  score on a scale | 50.9 (11.3)
Quality of Life (KOOS) [Mean (Standard Deviation); unit: score on a scale] — KOOS-QoL a self-reported measure consisting of 4 questions assessing quality of life, which is part of the five patient-relevant subscales of KOOS.The sub scale ranges from 0 to 100 where higher values represents a better outcome
  score on a scale | 27.4 (16.8)

OUTCOME MEASURES:

1. Primary Outcome: 30 Second Chair Standing Test
Description: The 30 second Chair Standing Test is one of three Osteoarthritis Research Society International (OARSI) recommended minimal core set of performance-based outcome measures in OA research and clinical practice.In this test, the subject will stand up completely from the sitting position so hips and knees are fully extended, then completely back in the seated position. This will be repeated for 30 seconds and the total number of chair stands will be recorded (up and down equals one stand).
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: stands
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
stands | 9.5 (0.5)

2. Primary Outcome: 40m Fast Paced Walking Test (40m FPWT)
Description: The 40-meter fast paced walk test is one of the three Osteoarthritis Research Society International recommended minimal core set of performance-based outcome measures in OA research and clinical practice.The subjects will be timed to complete a 40 m track course.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
seconds | 35.9 (2.6)

3. Primary Outcome: Timed Stair Climb
Description: The stair climb test is one of the three Osteoarthritis Research Society International recommended minimal core set of performance-based outcome measures in OA research and clinical practice. The subject will be timed while ascending and descending 9 steps of stairs.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: seconds
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
seconds | 15.0 (1.4)

4. Secondary Outcome: KOOS-PS (Knee Osteoarthritis Outcome Score - Physical Function Short Form)
Description: KOOS-Physical Function (KOOS-PS) Short Form is a parsimonious measure of physical function derived from the KOOS, which is a self-reported outcome score. The KOOS-Physical Function Short Form ranges from 0 to 100 where higher values represents a worse outcome.
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
score on a scale | 70.0 (2.1)

5. Other Pre Specified Outcome: KOOS-QoL (Knee Osteoarthritis Outcome Score - Quality of Life)
Description: KOOS-QoL a self-reported measure consisting of 4 questions assessing quality of life, which is part of the five patient-relevant subscales of KOOS.The sub scale ranges from 0 to 100 where higher values represents a better outcome
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
score on a scale | 51.9 (3.4)

6. Other Pre Specified Outcome: NRS for Pain
Description: The Numeric Rating Scale for Pain (NRS for Pain) is a measure of pain intensity. The subject will rate their knee pain bilaterally on a scale from no pain (0) to worst pain imaginable (10).
Time Frame: 12 weeks
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Intra-articular Zilretta Injection
Number analyzed (Participants) | 65
units on a scale | 3.3 (0.3)

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | Intra-articular Zilretta Injection
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 34/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intra-articular Zilretta Injection (N=70)
Allergic rhinitis (Immune system disorders) | 1 (1)
arthralgia (Musculoskeletal and connective tissue disorders) | 7 (7)
Blister (Skin and subcutaneous tissue disorders) | 1 (1)
Bruising (Blood and lymphatic system disorders) | 3 (3)
Epistaxis (Blood and lymphatic system disorders) | 1 (1)
Fall (General disorders) | 8 (8)
Flu-like symptoms (General disorders) | 1 (1)
headache (General disorders) | 2 (2)
Hematuria (Blood and lymphatic system disorders) | 1 (1)
Hyperglycemia (Endocrine disorders) | 1 (1)
Otitis media (Ear and labyrinth disorders) | 1 (1)
Rhinorrea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Swelling (Blood and lymphatic system disorders) | 2 (2)
URI (Renal and urinary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/40/NCT03895840/Prot_SAP_000.pdf